CLINICAL TRIAL: NCT05223712
Title: Artificial Intelligence System for the Detection and Prediction of Kidney Diseases Using Ocular Information
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: AIKD-2021
Record Dates: First submitted 2022-01-23; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Artificial Intelligence; Ophthalmology; Kidney Diseases
Keywords: Kidney Diseases; Artificial Intelligence; Eye information
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, urine and renal biopsy samples from CKD patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Development Dataset 01: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Department of Nephrology of the First Affiliated Hospital of Sun Yat-sen University
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases
- Development Dataset 02: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Medical Centre of Aikang Health Care, Guangzhou, China
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases
- Validation Dataset 01: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Department of Nephrology of the First Affiliated Hospital of Sun Yat-sen University
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases
- Validation Dataset 02: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Medical Centre of Aikang Health Care, Guangzhou, China
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases
- Test Dataset 01: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Department of Nephrology of the First Affiliated Hospital of Sun Yat-sen University
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases
- Test Dataset 02: Slit-lamp, retinal fundus images, OCTA and kidney diseases examinations collected from Medical Centre of Aikang Health Care, Guangzhou, China
  Interventions: Other: Diagnostic Test: Chronic Kidney Diseases

INTERVENTIONS:
Other: Diagnostic Test: Chronic Kidney Diseases — The development datasets were used to train the deep learning model, which was validated and tested by the other 4 datasets.

SUMMARY:
This is an retrospective and prospective multicenter study to develop and validate an artificial intelligent (AI) aided diagnosis, therapeutic effect assessment model including chronic kidney disease (CKD) and dialysis patients starting from April 2009, which is based on ophthalmic examinations (e.g. retinal fundus photography, slit-lamp images, OCTA, etc.) and CKD diagnostic and therapeutic data (routine clinical evaluations and laboratory data), to provide a reliable basis and guideline for clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously received kidney biopsy, ophthalmic examinations and routine examinations of the department of nephrology during in-hospital period with BCVA>0.5.

Exclusion Criteria:

* Patients without retinal fundus images or kidney diseases.
* The quality of the retinal fundus images can not meet the requirement for furthur analysis.
* Severe loss of results of routine examinations of the department of nephrology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who had slit-lamp, retinal fundus photography and kidney disease tests at the Department of Nephrology, First Affiliated Hospital of Sun Yat-sen University and Medical Centre of Aikang Health Care, Guangzhou, China
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-08-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve of the deep learning system | baseline
  The investigators will calculate the area under the receiver operating characteristic curve of deep learning system and compare this index between deep learning system and human doctors

SECONDARY OUTCOMES:
Sensitivity and specificity of the deep learning system | baseline
  The investigators will calculate the sensitivity and specifity of deep learning system and compare this index between deep learning system and human doctors

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No